CLINICAL TRIAL: NCT03640858
Title: Interventional Study to Assess the Effect of Expanded Dialysis Using the Theranova Dialyzer on Patient Reported Symptoms Using the London Evaluation of Illness (LEVIL)
Brief Title: Effect of Expanded Dialysis on Patient Reported Symptoms Using LEVIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics and Paediatrics, Robert Lindsay Chair of Dialysis Research and Innovation, London Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1589
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-03

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Larger middle molecules; Theranova
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Study visits take place within the patients' usual hemodialysis unit consistent with their routinely scheduled dialysis sessions. Beginning week 5 and 25 participants use the Theranova dialyzer until the end of the dialysis week on week 16 and 48. Participants answer 9 questions at least at one session regarding symptoms experienced since their last session using the LEVIL application. Furthermore, participants answer a single time to recovery question at the first treatment of weeks 1, 16, 24, and 48 to get more detailed information on recovery time after dialysis in addition to completing the 5-D Pruritus and the Restless Legs Syndrome scales.
  Bloodwork is drawn at 4 intervals throughout the study for laboratory evaluation.
  Participants have an echo at baseline and between weeks 12 to 16, 20-24 and 44-48 while on the Theranova dialyzer.
  In addition to this, participants will have non-invasive monitoring of circulatory stress using the CVInsight contact device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving hemodialysis (Experimental): A group of hemodialysis patients will be receiving the Theranova dialyzer during their regularly scheduled sessions to remove larger middle molecules
  Interventions: Device: Theranova Dialyzer

INTERVENTIONS:
Device: Theranova Dialyzer — The Theranova dialyzer will be used for each of the hemodialysis treatments beginning week 3 and ending at the end of the dialysis week on week 14 and again starting week 23 and ending at the end of the dialysis week on week 46 . This will allow us to compare patient reported symptoms in weeks 1 and 2 when patients are on their usual dialyzer with their symptoms using the Theranova dialyzer. This will also allow us to see if there is a carry-over effect.

SUMMARY:
Investigators know that many patients who are on dialysis suffer from the burden of unwanted symptoms, which can affect quality of life. In this study, the investigators will be assessing symptom burden using the London Evaluation of Illness "LEVIL," an application based platform where patients self-report their symptoms with at least one hemodialysis treatment. The investigators would like to compare the currently available dialyzer with a new dialyzer that is capable of removing solutes of higher molecular weight that may or may not cause patients to experience symptoms related to increased amounts of these toxins in their blood.

DETAILED DESCRIPTION:
Baxter Canada has an expanded hemodialysis (HDx) membrane called the "Theranova", which is capable of removing solutes of higher molecular weight. Although this clearly has biochemical advantages it is not known at this time if the removal of larger middle molecules can have a direct and immediate effect on patients reported symptoms and quality of life. In short, do be people actually feel better?

Given the way many QoL measurements fluctuate around the dialysis week, the investigators propose to utilize a dynamic tool. The investigators will be assessing symptom burden using the London Evaluation of Illness "LEVIL" an application based platform where patients self-report their symptoms with at least one hemodialysis treatment. Reports are generated immediately and in real-time, which cannot be accomplished with other symptom management tools. This allows the investigators to track study changes and benchmark observations to previously established baseline values. The investigators are excited to see if there is an imminent effect on how patients feel using the Theranova dialyzer.

The study is investigator initiated and the principal investigator has secured modest funding from Baxter to allow support for the core study team and the introduction and maintenance of the LEVIL evaluation platform at other centers. Baxter have also provided some dialyzer support, and will work with individual centers to ensure that there is no consumable increment of cost associated with participation.

The study is 60 weeks in length:

* LEVIL entries with at least one hemodialysis treatment each week for 60 weeks
* Blood sampling at 4 time points for all participants
* Implementation of Theranova dialyzer from weeks 5 through 16 and weeks 25 through 48
* Wash out period from weeks 17 through 24 and weeks 49 through 60
* Time to recovery question at the first treatment of weeks 1, 16, 24, and 48 for new participants
* 5-D Pruritus scale and Restless Legs Syndrome rating scale at the first treatment of weeks 1, 16, 24, and 48
* Echocardiogram prior to starting hemodialysis and at peak stress at baseline (within the first two weeks), with one treatment between weeks 12 to 16 which will occur mid-week, and with one treatment between weeks 44 to 48 which will occur mid-week (LHSC specific)
* CVInsight monitoring at baseline (within the first two weeks), with one treatment between weeks 2 to 16, 20 to 25, and with one treatment between weeks 44 to 48 (LHSC specific)
* Non-invasive assessment of cardiovascular risk using the AGE Reader within 1 hour of starting hemodialysis at baseline, with one treatment between weeks 12 to 16, 20 to 24, and with one treatment between weeks 44 to 48 which will occur mid-week (LHSC specific)
* Five Time Sit to Stand Test & 60-Second Chair Test at the second treatment of weeks 1, 16, 24, and 48

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patient
* Must be on hemodialysis for at least 3 months
* Age ≥18 years
* Willing and able to give informed consent

Exclusion Criteria:

* Active infection
* Active cancer
* Life expectancy <1 year as estimated by care provider
* Hemodialysis patients currently receiving Hemodiafiltration (HDF), Hemofiltration (HF) or Isolated ultrafiltration (ISO UF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
A change in larger middle molecule induced symptoms as assessed by the LEVIL application | Beginning week 1 and ending at the end of the dialysis week on week 46
  The primary outcome will be a change (from patient's own baseline) in general well-being, pain, sleep, breathing, energy, appetite, itch, restless legs, and recovery from hemodialysis when using the Theranova dialyzer. These parameters will be measured using the LEVIL an electronic application based visual analog scale.

SECONDARY OUTCOMES:
A change in larger middle molecule clearance using the Theranova dialyzer | First treatment of weeks 1, 14, and 46
  The secondary outcome is a change in the clearance of large middle molecules which will be evaluated by measuring levels of beta-2 microglobulin, beta-12 binding globulin, free light chains (kappa, lambda), factor D, fibroblast growth factor 23, and interleukin 6.
Correlation between large middle molecules and patient symptoms | Beginning week 1 and ending at the end of the dialysis week on week 54
  Another secondary outcome is the relationship between the clearance of large middle molecules and specific symptoms reported by the patients using the LEVIL application.
A change in symptoms with a change in dialyzer (usual to Theranova and vice versa) | Beginning week 1 and ending at the end of the dialysis week on week 54
  Another secondary outcome is if the time point where symptoms change with a change in dialyzer
Effect on microcirculation and/or hemodialysis induced circulatory stress with the Theranova dialyzer | Beginning week 3 and ending at the end of the dialysis week on week 14 and again week 23 and ending week 46
  Another secondary outcome is the Theranova dialyzer effect on microcirculation and/or hemodialysis induced circulatory stress

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McIntyre, MBBS DM, Principal Investigator — London Health Sciences Centre
Locations (2):
- Canada (2):
  - Adam Linton Dialysis Unit, London, Ontario
  - Kidney Care Centre, London, Ontario

REFERENCES:
- [Derived] Penny JD, Jarosz P, Salerno FR, Lemoine S, McIntyre CW. Impact of Expanded Hemodialysis Using Medium Cut-off Dialyzer on Quality of Life: Application of Dynamic Patient-Reported Outcome Measurement Tool. Kidney Med. 2021 Jul 29;3(6):992-1002.e1. doi: 10.1016/j.xkme.2021.05.010. eCollection 2021 Nov-Dec. PMID 34939008